CLINICAL TRIAL: NCT05154669
Title: Integrating Financial Coaching and Smoking Cessation Coaching for People With Low Income Who Smoke: a Randomized Controlled Trial
Brief Title: Integrating Financial Coaching and Smoking Cessation Coaching
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-00986; 1R01CA252483-01A1 (Other Grant/Funding Number: National Cancer Institute)
Record Dates: First submitted 2021-11-30; First posted 2021-12-13 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard Smoking Cessation Coaching (Active Comparator): Participants will receive 5 counseling sessions over approximately 8 weeks as per standard smoking cessation programs. Participants will receive 8 weeks of nicotine replacement therapy (patches, gum, and/or lozenges).
  Interventions: Drug: Nicotine Replacement Therapy Agent - Patches; Drug: Nicotine Replacement Therapy Agent - Lozenges; Drug: Nicotine Replacement Therapy Agent - Gum
- Integrated Financial-Smoking Cessation Coaching (Experimental): The integrated intervention will provide 5 counseling sessions over approximately 8 weeks that integrates financial coaching into the smoking cessation program. Participants will receive 8 weeks of nicotine replacement therapy (patches, gum, and/or lozenges).
  Interventions: Other: Financial counseling; Drug: Nicotine Replacement Therapy Agent - Patches; Drug: Nicotine Replacement Therapy Agent - Lozenges; Drug: Nicotine Replacement Therapy Agent - Gum

INTERVENTIONS:
Other: Financial counseling — The goals of the financial counseling will be to: (1) screen and refer participants to financial benefits and empowerment programs; (2) help participants create and maintain a household budget to meet short- and long-term goals; and (3) help participants link smoking cessation to their budgeting goals.
  Arms: Integrated Financial-Smoking Cessation Coaching
Drug: Nicotine Replacement Therapy Agent - Patches — 24 hour dosing system that provides regular, measured nicotine to the bloodstream through the skin. Nicotine patches are available in 3 dosages: 21 mg, 14mg, and 7mg. Patches will be adjusted based on withdrawal symptoms, urges, and comfort. After 4-6 weeks of abstinence, taper ever 2-4 weeks in 7-14 mg steps as tolerated.
Drug: Nicotine Replacement Therapy Agent - Lozenges — General Info 24 hour dosing system that provides regular, measured nicotine to the bloodstream through the skin.
  Provides regular, measured, amount of nicotine to the bloodstream through the mucous membranes of the mouth. As with the patch, the idea is to taper the amount of lozenges used until you no longer need it. Provides regular, measured, amount of nicotine to the bloodstream through the mucous membranes of the mouth. As with the patch and lozenge, the idea is to taper the amount of gum chewed until you no longer need it. Comes in 4mg or 2mg. Initial dosing is 1-2 lozenges every 1-2 hours (minimum of 9/day). Taper as tolerated
Drug: Nicotine Replacement Therapy Agent - Gum — Provides regular, measured, amount of nicotine to the bloodstream through the mucous membranes of the mouth. As with the patch and lozenge, the idea is to taper the amount of gum chewed until you no longer need it. Initial dosing is 1-2 pieces every 1-2 hours (10-12 pieces/day). Taper as tolerated

SUMMARY:
This study conduct a two-arm, parallel-group randomized controlled trial. The study will recruit and randomize 900 smokers (n=450 per arm) to either: (1) Control: Standard Smoking Cessation Counseling or (2) Intervention: Integrated Financial-Smoking Cessation Counseling.

DETAILED DESCRIPTION:
The study is a two-arm, parallel-group RCT. The study will recruit and randomize 900 low-income smokers (n=450 per arm) to either: (1) Control: Standard Smoking Cessation Counseling or (2) Intervention: Integrated Financial-Smoking Cessation Counseling. Both groups will receive 8 weeks of nicotine replacement therapy. The study will survey participants at baseline, 6 months, and 12 months to assess outcomes and mechanisms, and biochemically verify self-reported abstinence at 12 months (our primary outcome). The study will assess and compare the costs and cost-per-quit in the two treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years,
* smokes ≥5 cigarettes per day,
* interested in receiving smoking and financial counseling,
* self-reported income below 200% of the current federal poverty level,
* New York City resident,
* speaks English or Spanish language (the interventions and measures have not been validated in other languages),
* able to provide informed consent, and
* does not have a representative who manages his/her funds.

Exclusion Criteria

* people who know a current past study participant (to avoid intervention contamination)
* People who have a medical contraindication to using nicotine replacement therapy:
* allergy to nicotine patch
* pregnancy or intention to become pregnant over the next 12 months
* breastfeeding
* heart attack in the past 2 months
* underlying arrhythmia
* ongoing or worsening angina.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 488 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the integrated intervention to standard cessation counseling on long-term abstinence (salivary cotinine) | 12 months
  The study will collect salivary cotinine from participants reporting 7-day abstinence from cigarettes on the 12-month survey. The study will use a saliva collection kit supplied by Salimetrics Inc. Participants will be classified as negative for salivary cotinine if their concentration is <10ng/ml,
Effectiveness of the integrated intervention to standard cessation counseling on long-term abstinence (CO concentration) | 12 months
  The study will collect exhaled CO from participants reporting 7-day abstinence from cigarettes on the 12-month survey. The study will use a coVita Co monitor that provides an immediate CO concentration reading in single parts per million (ppm). Participants will be classified as negative for exhaled CO if their concentration is <8 ppm.

SECONDARY OUTCOMES:
Change in quit attempts | 6 and 12 months
  Measured with self reported survey regarding attempts to quit smoking at 6 months and at 12 months
Change in self-reported abstinence from cigarettes | 6 and 12 months
  Measured with self-reported abstinence from cigarettes at 6 months and at 12 months
Change in self-reported use of electronic nicotine delivery systems use | 6 and 12 months
  Measured with self-reported use of electronic nicotine delivery systems use at 6 months and at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Erin Rogers, DrPH, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to ERIN.ROGERS@NYULANGONE.ORG. To gain access, data requestors will need to sign a data access agreement.